CLINICAL TRIAL: NCT07128966
Title: Joined Bio - JB-MR-250225, Direct to Patient Minimal Risk Research
Brief Title: Direct to Patient Minimal Risk Biospecimen and Data Collection Research
Acronym: JBMR
Status: Not yet recruiting | Type: Observational
Sponsor: Joined Bio (Industry)
Responsible Party: Sponsor
Other Study IDs: JB-MR-250225; JB Direct to Participant (Other: Joined Bio)
Record Dates: First submitted 2025-08-11; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Healthy; Lupus; Celiac; Kidney Disease; Chronic; Dermatologic
Keywords: biospecimen; rare disease; participant
MeSH Terms: conditions — Celiac Disease; Kidney Diseases; Bronchiolitis Obliterans Syndrome; Rare Diseases | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Minimal risk only:
  Blood hair, nail, skin scrapings urine, stool, sweat, tears uncannulated saliva; mucosal and skin cells collected by buccal scraping or mouth washings; sputum collected after saline mist nebulization; nasal swabs that are inserted no deeper than until resistance is met (i.e. are not inserted beyond the opening of the nasal cavity into the pharynx); cheek or throat swabs; vaginal swabs when no deeper than 4 inches or until resistance is met (i.e. do not go beyond the opening to the cervix); external genital swabs.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy participants: This is non-interventional, observational only research. Participants may be healthy. Participants will be invited to participate on a per-project basis, depending on the cohort requirements for the project.
  Interventions: Other: Observation
- Participants with a condition: Participants may have a condition such as lupus, celiac, dermatitis or other condition. Participants will be invited to participate on a per-project basis, depending on the cohort requirements for the project.
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — This is non-interventional, observational only

SUMMARY:
This study aims to help researchers better understand health conditions and develop improved tests, treatments, and cures for diseases. Joined Bio collects health data, lifestyle information, biological samples, and feedback from participants and provides this to qualified research partners.

DETAILED DESCRIPTION:
Primary: The primary objective of this study is to connect participants with specific health profiles, along with biospecimens and associated de-identified health data, to scientific researchers who are searching for new diagnostics and treatments for a wide array of conditions. This will accelerate medical discovery by connecting medical research with the power of patient participation.

Secondary: The secondary objective of this study is to allow participants with specific health profiles, along with their de-identified health data, to help further the cause of medicine generally through interviews, surveys, and other minimal risk research activities desired by life science organizations.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, that are adults [have reached the Age of Majority = aged 18 to 90 in most US states; aged 19-90 in Alabama or Nebraska; aged 21-90 in Mississippi or Puerto Rico].
* Have reviewed and signed a consent or e-consent form for this study. If a person with diminished decision-making capacity, their Legally Authorized Representative has reviewed and signed the consent for on their behalf.
* Be willing to comply with all study procedures and be available for the duration of the study.
* Meets requirements of a current request for research participation (e.g. has previous diagnosis of a medical condition of interest or laboratory results within a specific range).
* Pregnant women may be enrolled in this study in accordance with 45 CFR Part 46 Subpart B.

Exclusion Criteria:

* Unable to meet the Inclusion Criteria listed above.
* Prisoners or children
* Unable to provide the requested biospecimen(s), data or feedback without placing the individual at risk.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Outside of this protocol, Joined Bio is creating a network of individuals who are interested in participating in research. Individuals are recruited across a broad cross-section of ages, medical conditions, and geographic locations within the United States. These individuals voluntarily join the Joined Bio network, consent to share health information with Joined, and then securely transfer their health information to Joined Bio. All health information is stored in a de-identified manner (with the exception of dates of service, which are protected in accordance with HIPAA) and encrypted with Joined Bio holding re-identification keys.
  Joined Bio then searches its network of participants to see if there are matches to the research project. If there are matches, Joined Bio re-identifies the individual and reaches out to them to let them know that they match up to a research project and also to provide them with information about the research.
Sampling Method: Non-Probability Sample
Enrollment: 100000 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2035-09-01 (Estimated); Study Completion 2036-09-01 (Estimated)

PRIMARY OUTCOMES:
Observation for biomarker identification | 10 years
  There is no defined study outcome. Rather this is an observational study of multiple participant populations that hopes to identify new biomarkers, treatments and/or diagnostic applications.

CONTACTS AND LOCATIONS:
Overall Officials: Chris Ianelli, MD, Principal Investigator — Joined Bio
Locations (1):
- Joined Bio, Lexington, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://joined.bio/